CLINICAL TRIAL: NCT01292564
Title: An Evaluation of the Effect of the Erchonia ML Scanner (MLS) as Applied to Body Contouring of the Waist and Hips on Fat Emulsification Pilot Study.
Brief Title: Study to See How Low Level Laser Light Affects Subcutaneous Fat Around the Hips and Waist
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient resources at test site for recruitment.
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EC-MRI001
Record Dates: First submitted 2011-02-08; First posted 2011-02-09 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Erchonia MLS (Active Comparator): The Erchonia MLS emits 635 nm low level laser light.
  Interventions: Device: Erchonia MLS
- Placebo Laser (Placebo Comparator): The Placebo Laser looks identical to the Erchonia MLS Laser but emits no therapeutic light.
  Interventions: Device: Placebo Laser

INTERVENTIONS:
Device: Erchonia MLS — The Erchonia MLS emits 635 nm low level laser light.
  Arms: Erchonia MLS
Device: Placebo Laser — The Placebo Laser looks identical to the Erchonia MLS Laser but emits no therapeutic light.
  Arms: Placebo Laser

SUMMARY:
The purpose of this pilot study is to demonstrate the anatomical modulation of subcutaneous fat across the waist and hips that occurs through application of the Erchonia® ML Scanner (MLS) Laser manufactured for non-invasive body contouring of the waist and hips.

DETAILED DESCRIPTION:
Laser therapy provides an alternative therapeutic regimen for the reduction of subcutaneous tissue volume. Although the biochemical mechanism is not yet fully understood, histological studies clearly and effectively identify the formation of the transitory pore and subsequent cell collapse immediately following laser irradiation. More importantly, a placebo-controlled, randomized, double-blind clinical investigation using the Erchonia MLS with 67 enrolled participants revealed a statistically significant reduction of overall circumference measurements of the waist, hip, and thighs following two weeks of treatment, resulting in Food and Drug Administration (FDA) clearance for the indication.

Laser therapy operates under the principle of photochemistry, activating and/or suppressing natural biochemical processes. Because Low Level Laser Therapy (LLLT) does not induce cellular apoptosis, there is no upregulation of pro-inflammatory cytokines nor is there a large burden placed on the lymphatic system. The fatty material secreted from the adipocytes following laser irradiation are absorbed by the lymphatic system, broken down by the liver, and naturally secreted. Fatty acids released are bound to albumin, and are transported through the circulatory system to the liver to undergo fatty acid oxidation. The triglycerides released are bound as lipoproteins and transported to the liver to be processed. Moreover, a lipase known as lipoprotein lipase, has been demonstrated to breakdown emulsified triglycerides; therefore breaking the molecule down into three fatty acids and one glycerol molecule. The most important aspect of laser therapy is that cellular apoptosis is not induced. The fatty material being evacuated from the cell must be absorbed by the lymphatic system, and because laser therapy does not destroy the cell, the complex organelles and the entire cell structure will not be absorbed by the lymphatic system. It is not well understood how much the lymphatic system can absorb; therefore, creating a mass amount of cellular debris by destroying adipose tissue may result in serious long term effects. Moreover, adipose tissue is not just composed of fat storing cells; there is also a collection of immune cells, fibroblasts, vessels, and stromal stem cells. By creating the transitory pore in the fat storing cell only, the viability of the surrounding, non-fat storing cells is preserved.

The purpose of this pilot study is to demonstrate and document the anatomical modulation of subcutaneous fat across the waist and hips that occurs through application of the Erchonia® ML Scanner (MLS) Laser manufactured for non-invasive body contouring of the waist and hips.

ELIGIBILITY:
Inclusion Criteria:

* Subject indicated for liposuction or use of liposuction techniques for the removal of localized deposits of adipose tissues; specifically for the indication of body contouring in the areas of the waist and hips. (As per the American Academy of Cosmetic Surgery's 2006 Guidelines for Liposuction Surgery).
* Body Mass Index (BMI) of 28 to 43 kg/m², inclusive.
* It is deemed safe for the subject to undergo a MRI procedure based on the MRI screening questionnaire.
* Subject is willing and able to abstain from partaking in any treatment other than the study procedure to promote body contouring and/or weight loss during study participation.
* Subject is willing and able to maintain his or her regular diet and exercise regimen without effecting significant change in either direction during study participation.

Exclusion Criteria:

* Body Mass Index (BMI) is less than 28 kg/m² or greater than 43 kg/m².
* Diabetes dependent on insulin or oral hypoglycemic medications.
* Known cardiovascular disease.
* Prior cardiac surgery.
* Prior surgical intervention for body sculpting/weight loss.
* Medical, physical, or other contraindications for body sculpting/weight loss.
* Current use of medication(s) known to affect weight levels/bloating/swelling and for which abstinence during study participation is not safe or medically prudent.
* Any medical condition known to affect weight levels/cause bloating/swelling.
* Diagnosis of, and/or taking medication for, irritable bowel syndrome.
* Active infection, wound or other external trauma to the laser treatment area.
* Pregnant, breast feeding, or planning pregnancy prior to study end.
* Serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in past two years.
* Developmental disability or cognitive impairment that would preclude adequate comprehension of the informed consent form and/or ability to record study measurements.
* Involvement in litigation and/or a worker's compensation claim and/or receiving disability benefits related to weight-related and/or body shape issues.
* participation in research in the past 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Fat Surface area (cm2) & projected fat volume (cm3) determined through MRI analysis | 2 weeks

SECONDARY OUTCOMES:
Body Mass Index (BMI) | 2 weeks
Hip circumference measurement in cm | 2 weeks
Waist circumference measurement | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Turok, MD, Principal Investigator
Locations (1):
- American Laser Centers, Fox River Grove, Illinois, United States